CLINICAL TRIAL: NCT02357888
Title: Double-blind, Randomized, Placebo-controlled, Cross-over Study of the Effect of a 2.5 mg Nicotine Lozenge on Smoking Craving
Brief Title: Assessment of V0018 2.5 mg Effect on Craving
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pierre Fabre Medicament (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: V00018 PC 2 06; 2014-004387-38 (EudraCT Number)
Record Dates: First submitted 2015-02-03; First posted 2015-02-06 (Estimated); Last update posted 2015-10-08 (Estimated); Status verified 2015-10

CONDITIONS: Healthy Highly Dependant Smokers
Keywords: Nicotine replacement therapy; craving

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Sequence 1 (Experimental): Treatment group sequence: Test Product on Day 1 and Placebo on Day 2
  Interventions: Drug: V0018; Drug: Placebo
- Sequence 2 (Experimental): Treatment group sequence: Placebo on Day 1 and Test Product on Day 2
  Interventions: Drug: V0018; Drug: Placebo

INTERVENTIONS:
Drug: V0018 — Oromucosal - Single dose
Drug: Placebo — Oromucosal - Single dose

SUMMARY:
The purpose of this study is to evaluate the reduction of craving and its time course after administration of V0018 2.5 mg compared to placebo in healthy highly dependant smokers.

ELIGIBILITY:
Inclusion Criteria:

* Male and female aged 18 to 64 years
* Smoking ≥ 20 cigarettes/day continuously for the last two years
* With a first cigarette smoked within 30 min after waking
* Not currently in the process of quitting smoking

Exclusion Criteria:

Related to pathologies

* Current or recurrent buccal lesions which, in the opinion of the investigator, would interfere with the assessment of the different parameters
* Hyposalivation or asialia
* Intolerance to lactose, or any pathology that could cause endogenous production of carbon monoxide (CO)

Related to treatments

* Use of antidepressants within the last three months
* Use of sedatives, hypnotics, tranquilizers or any other addictive agents within the last 3 months
* Routine use of tobacco other than cigarettes
* Regular use for more than one week of any treatment for smoking cessation (gum, patch, inhaler, lozenge, tablet, bupropion, varenicline) and other smokeless tobacco products (including e-cigarettes) within three months
* History of hypersensitivity to nicotine, peanut, soya or to any of the excipients of study treatment
* Intolerance to fructose
* History of phenylketonuria (aspartame)

For women of childbearing potential:

* Is pregnant or in post-partum period or a nursing mother

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2015-02; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Questionnaire for Smoking Urges Brief (QSU-Brief) (10 items) | 15 minutes
  Change from study baseline to 15 minutes after treatment intake for the QSU-brief total score and demonstrate any earlier effect.

CONTACTS AND LOCATIONS:
Overall Officials: Françoise MD TONNER, Study Director — Pierre Fabre Medicament
Locations (1):
- Gières, France